CLINICAL TRIAL: NCT01353287
Title: Transcatheter Aortic Valve Intervention-Live Transmission (VERITAS)Study
Brief Title: Transcatheter Aortic Valve Intervention-Live Transmission
Acronym: VERITAS
Status: Completed | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: VERITAS
Record Dates: First submitted 2011-05-11; First posted 2011-05-13 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Aortic Valve Disorder
Keywords: Transcatheter Aortic Valve Intervention (TAVI); Live case transmission
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- TAVI live case or video-taped transmission
- TAVI without transmission

SUMMARY:
The primary objective of this clinical trial is to evaluate safety of patients who underwent Transcatheter Aortic Valve Intervention (TAVI) during a live case or video-taped transmission as compared to those without procedure transmission.

DETAILED DESCRIPTION:
A series of sites from outside the US, where the Edwards-Sapien and CoreValve devices are approved for commercial sale and implantation, will be recruited to retrospectively identify and extract in-hospital data of a patient who underwent TAVI during a live or video-taped procedure and a matched patient who underwent TAVI without transmission of the procedure.

ELIGIBILITY:
Cases Inclusion Criteria:

* Subjects > 18 years of age, male or female
* Subject had live case or video-taped transmission of TAVI procedure with:

Edwards-Sapien transfemoral approach, Edwards-Sapien transapical approach, or CoreValve transfemoral approach

Controls Inclusion Criteria:

* Subjects > 18 years of age, male or female
* Subject underwent TAVI without procedure transmission and had:

Edwards-Sapien transfemoral approach, Edwards-Sapien transapical approach, or CoreValve transfemoral approach

* Subjects will be matched to Cases upon the following:
* STS SCORE +/- 2points
* Date of TAVI procedure +/- 4weeks
* The first attending for the TAVI procedure
* Access site for TAVI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, male or female, over 18 years of age who have either undergone live case or video-taped transmission of TAVI procedure (Case), or have undergone the procedure without procedure transmission(Control).
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2011-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Major complication defined as in hospital death, stroke, tamponade, valve embolization, coronary obstruction, renal failure requiring dialysis, and the need for a pacemaker. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Washington Hospital Center, Washington, DC
Locations (6):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States
- Saint Paul's Hospital, Vancouver, British Columbia, Canada
- CardioVasculares Centrum Frankfurt, Frankfurt, Germany
- San Raffaele Hospital, Milan, Italy
- Bern University Hospital, Bern, Switzerland
- Guys and St Thomas' Hospital, London, United Kingdom